CLINICAL TRIAL: NCT00097084
Title: Efficacy and Safety Comparison of Insulin Detemir Plus Insulin Aspart Versus Insulin Glargine Plus Insulin Aspart in Type 2 Diabetes
Brief Title: Comparison of Insulin Detemir Plus Insulin Aspart Against Insulin Glargine Plus Insulin Aspart in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1431; 2004-000087-27 (EudraCT Number)
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin glargine
Drug: insulin aspart

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The purpose of this study is to test whether insulin detemir is a safe and at least as effective alternative to insulin glargine for the control of blood glucose in basal/bolus therapy in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months
* Treated with oral antidiabetic drugs or with any insulin regimen with or without oral antidiabetic drugs
* BMI of maximum 40 kg/m2
* HbA1c greater than or equal to 7.0% and less than or equal to 11.0%

Exclusion Criteria:

* Proliferative retinopathy or maculopathy
* Recurrent major hypoglycaemia
* Impaired hepatic or renal function
* Cardiac problems or uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2004-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 1 year trial period

SECONDARY OUTCOMES:
Adverse events
Body weight
Hypoglycemia
Blood glucose
Insulin Treatment Satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (57):
- United States (26):
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, San Francisco, California
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Lake Mary, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Palm Harbor, Florida
  - Novo Nordisk Investigational Site, Vero Beach, Florida
  - Novo Nordisk Investigational Site, Athens, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Berlin, New Jersey
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Hermitage, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Tacoma, Washington
- Finland (7):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kurikka
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Lapua
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Turku
- France (9):
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Le Mans
  - Novo Nordisk Investigational Site, Montpellier
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Narbonne
  - Novo Nordisk Investigational Site, Nevers
  - Novo Nordisk Investigational Site, Orléans
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Vénissieux
- Norway (6):
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Notodden
  - Novo Nordisk Investigational Site, Sarpsborg
  - Novo Nordisk Investigational Site, Ski
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- Sweden (9):
  - Novo Nordisk Investigational Site, Ängelholm
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Kalmar
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Motala
  - Novo Nordisk Investigational Site, Oskarshamn
  - Novo Nordisk Investigational Site, Uddevalla

REFERENCES:
- [Result] Hollander P, Cooper J, Bregnhoj J, Pedersen CB. A 52-week, multinational, open-label, parallel-group, noninferiority, treat-to-target trial comparing insulin detemir with insulin glargine in a basal-bolus regimen with mealtime insulin aspart in patients with type 2 diabetes. Clin Ther. 2008 Nov;30(11):1976-87. doi: 10.1016/j.clinthera.2008.11.001. PMID 19108786
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com